CLINICAL TRIAL: NCT06984458
Title: Exploring the Impact of Dementia Prevention Programs Using Robots as Intervention Tools on Community Elderly
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202503HM004
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia; Cognitive Decline; Psychological Well-being; Aging and Cognitive Health
Keywords: Robot-delivery intervention, Dementia prevention, Dementia, Community elderly
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dementia Prevention Programs Using Robots as Intervention Tools (Experimental): The experimental group conducted a two-month "Robot Dementia Prevention Course" intervention. The research subjects were 40 people. Each group of 5 people was assigned a Kebbi robot. The course intervention was divided into 8 groups. The Kebbi robot mainly taught and communicated with the elderly interactively. There is a well-trained teaching assistant in the class to enhance the learning effect of the elderly. The two classes per week are about 2 hours long, with 50 minutes of course knowledge introduction, 10 minutes of rest, 50 minutes of interaction with Kebbi Artificial Intelligence-based board games, and 10 minutes of prize-based quizzes after class. They are held once a week, with a total of 8 weeks of courses (duration two months).
  Interventions: Behavioral: Robot Dementia Prevention Course
- Control group (No Intervention): The control group did not receive any course intervention. The community elderly were given a pre-test. After 8 weeks (two months), the f post-test will be conducted.

INTERVENTIONS:
Behavioral: Robot Dementia Prevention Course — It is expected that through the eight-week course design activities, the cognitive functions, social activities, emotional management (such as alleviating depression), well-being, reduce loneliness and can be achieved, thereby preventing or delaying cognitive decline.
  The experimental group conducted a two-month "Robot Dementia Prevention Course" intervention. The research subjects were 40 people. Each group of 5 people was assigned a Kebbi robot. The course intervention was divided into 8 groups. The Kebbi robot mainly taught and communicated with the elderly interactively. There is a well-trained teaching assistant in the class to enhance the learning effect of the elderly. The two classes per week are about 2 hours long, with 50 minutes of course knowledge introduction, 10 minutes of rest, 50 minutes of interaction with Kebbi Artificial Intelligence-based board games, and 10 minutes of prize-based quizzes after class.
  Arms: Dementia Prevention Programs Using Robots as Intervention Tools

SUMMARY:
The purpose of this study is to intervene in the cognitive functions of the community elderly through the "Robot Dementia Prevention Course" training. It is expected that through the eight-week course design activities, the cognitive functions, social activities, emotional management (such as alleviating depression), well-being, reduce loneliness and can be achieved, thereby preventing or delaying cognitive decline.

This study is a quasi-experimental design. It adopts pre-test and post-test methods for the experimental group and the control group. Before the intervention of the "Robotic Dementia Prevention Course", the community elderly were given a pre-test. After receiving an 8-week course (two months), the first post-test will be conducted, and three months later, the second post-test (post-post-test) will be conducted to analyze the delay effect. The experimental group conducted a two-month "Robot Dementia Prevention Course" intervention. The research subjects were 40 people. Each group of 5 people was assigned a Kebbi robot. The course intervention was divided into 8 groups. The Kebbi robot mainly taught and communicated with the elderly interactively. There is a well-trained teaching assistant in the class to enhance the learning effect of the elderly. The two classes per week are about 2 hours long, with 50 minutes of course knowledge introduction, 10 minutes of rest, 50 minutes of interaction with Kebbi Artificial Intelligence-based board games, and 10 minutes of prize-based quizzes after class. They are held once a week, with a total of 8 weeks of courses (duration two months), classes were taken in the elderly's original care center or long-term care base; the control group did not receive any course intervention. Statistical methods were analyzed using SPSS version 23.0, and descriptive statistics, paired t tests, generalized estimating equations, etc. were used to test the changes before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older, Able to communicate in Mandarin or Taiwanese, Able to provide informed consent or have a legal guardian provide consent

Exclusion Criteria:

* Diagnosis of severe dementia or advanced neurodegenerative disease, Severe psychiatric disorders (e.g., schizophrenia, bipolar disorder), Unconsciousness or inability to stay awake or focused for the session duration, Inability to comply with study protocol or scheduled sessions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-18 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function Assessed by SPMSQ | Participants will complete the SPMSQ at baseline, post-intervention (week 8), and follow-up (week 20).
Change in Depression Symptoms Assessed by GDS-15 | The instrument will be administered at baseline, post-intervention (week 8), and follow-up (week 20).
Change in Social Engagement and Activities Assessed by SEAQ | The instrument will be administered at baseline, post-intervention (week 8), and follow-up (week 20).
Change in Psychological Well-being Assessed by WHO-5 | The instrument will be administered at baseline, post-intervention (week 8), and follow-up (week 20).
Change in loneliness Assessed by UCLA Loneliness Scale | The instrument will be administered at baseline, post-intervention (week 8), and follow-up (week 20).

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Long Guo, PhD, Study Chair — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided